CLINICAL TRIAL: NCT05110716
Title: Effects of Choice Bundling on Valuation of Delayed Gains and Losses in Cigarette Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Minnesota (Other)
Responsible Party: Principal Investigator, Jeffrey Stein, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 20-827; 5P01CA217806 (NIH)
Record Dates: First submitted 2021-10-11; First posted 2021-11-08 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Cigarette Smoking
Keywords: Behavior; Smoking; Cigarette; Tobacco; Delay discounting; Intertemporal choice
MeSH Terms: conditions — Cigarette Smoking; Behavior; Smoking

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either a gains or losses group and subsequently complete conditions at bundle-sizes 1, 3, and 9 (within-subjects, order counterbalanced).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data collection and randomization to groups was performed online without the investigators' direct involvement
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Gains, Ascending Bundle-Size Order (Experimental): Participants will complete the choice bundling adjusting-amount task for monetary gains in an ascending order of bundle size.
  Interventions: Behavioral: Bundle-size 1; Behavioral: Bundle-size 3; Behavioral: Bundle-size 9
- Gains, Descending Bundle-Size Order (Experimental): Participants will complete the choice bundling adjusting-amount task for monetary gains in a descending order of bundle size.
  Interventions: Behavioral: Bundle-size 1; Behavioral: Bundle-size 3; Behavioral: Bundle-size 9
- Losses, Ascending Bundle-Size Order (Experimental): Participants will complete the choice bundling adjusting-amount task for monetary losses in an ascending order of bundle size.
  Interventions: Behavioral: Bundle-size 1; Behavioral: Bundle-size 3; Behavioral: Bundle-size 9
- Losses, Descending Bundle-Size Order (Experimental): Participants will complete the choice bundling adjusting-amount task for monetary losses in an ascending order of bundle size.
  Interventions: Behavioral: Bundle-size 1; Behavioral: Bundle-size 3; Behavioral: Bundle-size 9

INTERVENTIONS:
Behavioral: Bundle-size 1 — In this condition, each choice in the adjusting-amount task produces only a single consequence (e.g., lose $900 in 1 year).
Behavioral: Bundle-size 3 — In this condition, each choice in the adjusting-amount task produce a series of three consequences over time. o hold total amount constant across conditions, the $900 available in the bundle-size 1 condition will be distributed equally across all consequences in the series. (e.g., lose $300 in 1 year, lose $300 in 2 years, lose $300 in 3 years).
Behavioral: Bundle-size 9 — In this condition, each choice in the adjusting-amount task produce a series of nine consequences over time. To hold total amount constant across conditions, the $900 available in the bundle-size 1 condition will be distributed equally across all consequences in the series. (e.g., lose $100 in 1 year, lose $100 in 2 years, lose $100 in 3 years...lose $100 in 9 years).

SUMMARY:
The present study will investigate the effects of choice bundling, in which a single choice produces a series of repeating consequences, on valuation of delayed monetary gains and losses in an online panel of cigarette smokers.

DETAILED DESCRIPTION:
Choice bundling, in which a single choice produces a series of repeating consequences, has been shown to increase valuation of delayed monetary and non-monetary gains. Interventions derived from this manipulation may be an effective method for mitigating the elevated delay discounting rates observed in cigarette smokers. No prior work, however, has investigated whether effects of choice bundling generalize to reward losses. In the present study, an online panel of cigarette smokers, recruited using Ipsos, will complete assessments for either monetary gains or losses (randomly assigned). In Step 1, participants will complete a delay-discounting task to establish Effective Delay 50 (ED50), or the delay required for a monetary outcome to lose half of its value. In Step 2, participants will complete three conditions of an adjusting-amount task, choosing between a smaller, sooner (SS) adjusting amount and a larger, later (LL) fixed amount. The bundle size (i.e., number of consequences) will be manipulated across conditions, where a single choice will produce either 1 (control), 3, or 9 consequences over time (ascending/descending order counterbalanced). The delay to the first LL amount in each condition, as well as the intervals between all additional SS and LL amounts (where applicable), will be set to individual participants' ED50 values from Step 1 to control for differences in discounting of gains and losses.

ELIGIBILITY:
Inclusion Criteria:

* currently smoke at least 10 cigarettes per day
* have smoked at least 100 cigarettes (lifetime), and
* are 21 years of age or older.

Exclusion Criteria:

* Inaccurate identification of usual brand cigarette's as menthol or non-menthol

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
Indifference points | 1 day (same session)
  Participants complete three conditions of the adjusting-amount task (one at each bundle size), in which they choose between a larger, delayed amount ($900) and a smaller, immediate amount. Across trials, the smaller amount titrates until reaching an indifference point. This indifference point provides an index of the value of the larger option. For example, an indifference point of $300 indicates the larger, delayed amount as been discounted by two thirds. Higher values reflect less delay discounting.

CONTACTS AND LOCATIONS:
Overall Officials: Warren K Bickel, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be made available from the Open Science Framework (OSF) database. The url providing access to data will be provided in study publications.
Time Frame: Data will become available immediately upon publication of the manuscript and will remain available for 5 years.